CLINICAL TRIAL: NCT06704139
Title: Role of Prophylactic Antiemetics in Women Receiving Intrathecal Morphine and Lipophilic Opioids Added to Bupivacaine for Cesarean Section
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Maher Ywakim, resident doctor at anesthesia and ICU department Faculty of Medicine, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: antiemetics cesarean section
Record Dates: First submitted 2024-11-22; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Cesarean Section
Keywords: prophylactic antiemetics
MeSH Terms: interventions — Morphine; Fentanyl; Ondansetron; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be allocated in 1: 1 ratio into the two study groups using a web-based randomiser (https://www.randomizer.org/) to generate codes placed within sealed, opaque, sequentially numbered envelopes by a research assistant who will not be involved in patient care or assessment. This assistant also will prepare the study solutions in identical syringes that will be labelled ''study drug'' according to the assigned group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group 1 (Experimental): Fifty patients will receive intrathecal morphine
  Interventions: Drug: Morphine - .25 mg; Drug: Ondansetron + Dexamethasone
- group 2 (Experimental): Fifty patients will receive intrathecal morphine and fentanyl
  Interventions: Drug: fentanyl + morphine; Drug: Ondansetron + Dexamethasone

INTERVENTIONS:
Drug: Morphine - .25 mg — Fifty patients will receive intrathecal morphine
  Arms: group 1
Drug: fentanyl + morphine — Fifty patients will receive intrathecal morphine and fentanyl
  Arms: group 2
Drug: Ondansetron + Dexamethasone — All patients will receive a compination of intravenous 4mg ondansteron and 8mg dexamethasone 15 minutes before spinal anathesia

SUMMARY:
Because the majority of Caesarean deliveries are performed under neuraxial anaesthesia, Intrathecal morphine has become the gold standard for post-Caesarean delivery analgesia. However, postoperative nausea and vomiting (PONV) is the common side-effect of intrathecal morphine, affecting up to 60-80% of women without prophylaxis. PONV reduces maternal satisfaction and delays discharge from hospital, so it is important to prevent PONV in contemporary obstetric anaesthesia, particularly in the context of Enhanced Recovery After Surgery (ERAS) after Caesarean delivery.

According to the meta-analysis by Lizhong Wang et al., combined 5-HT3 antagonists plus dexamethasone are more effective than mono-therapy in preventing PONV associated with intrathecal morphine after Caesarean delivery. But, the role of prophylactic antiemetics in women receiving intrathecal morphine and lipophilic opioids is still unclear. As antiemetics were shown to be less effective in women receiving intrathecal morphine than in those receiving epidural morphine, Lizhong Wang et al., performed a further subgroup analysis based on whether intrathecal morphine was combined with lipophilic opioids or not. Surprisingly, the results in women who received intrathecal morphine alone were similar to those in the primary analyses; however, in those who received intrathecal morphine and lipophilic opioids, there were no statistical differences in almost all comparisons. This raises the question of whether the combination of intrathecal lipophilic opioids contributed to the reduced efficacy of antiemetics in women receiving intrathecal morphine The objective of the current study is to examine the effect of prophylactic use of combined 5-HT3 antagonists plus dexamethasone to decrease the incidence of postoperative nausea and vomiting in parturients undergoing CS under spinal anaesthesia who receive intrathecal morphine alone or combined with lipophilic opioids.

DETAILED DESCRIPTION:
Because the majority of Caesarean deliveries are performed under neuraxial anaesthesia, Intrathecal morphine has become the gold standard for post-Caesarean delivery analgesia. However, postoperative nausea and vomiting (PONV) is the common side-effect of intrathecal morphine, affecting up to 60-80% of women without prophylaxis. PONV reduces maternal satisfaction and delays discharge from hospital, so it is important to prevent PONV in contemporary obstetric anaesthesia, particularly in the context of Enhanced Recovery After Surgery (ERAS) after Caesarean delivery.

According to the meta-analysis by Lizhong Wang et al., combined 5-HT3 antagonists plus dexamethasone are more effective than mono-therapy in preventing PONV associated with intrathecal morphine after Caesarean delivery. But, the role of prophylactic antiemetics in women receiving intrathecal morphine and lipophilic opioids is still unclear. As antiemetics were shown to be less effective in women receiving intrathecal morphine than in those receiving epidural morphine, Lizhong Wang et al., performed a further subgroup analysis based on whether intrathecal morphine was combined with lipophilic opioids or not. Surprisingly, the results in women who received intrathecal morphine alone were similar to those in the primary analyses; however, in those who received intrathecal morphine and lipophilic opioids, there were no statistical differences in almost all comparisons. This raises the question of whether the combination of intrathecal lipophilic opioids contributed to the reduced efficacy of antiemetics in women receiving intrathecal morphine

ELIGIBILITY:
Inclusion Criteria:

* • Age from 19 to 40 years old.

  * Singleton pregnancies with a gestational age of at least 37 weeks.
  * pregnant women are scheduled for elective caesarean delivery.
  * Patients with stable vital signs.
  * Patients with normal laboratory investigations.
  * patients undergoing spinal anaesthesia for caesarean delivery via Pfannenstiel incision with exteriorization of the uterus

Exclusion Criteria:

* • Patient's refusal.

  * Age < 19 or > 40 years.
  * Height<150 cm, weight < 60 kg, body mass index (BMI) ≥40 kg/m2.
  * Contraindications to spinal anaesthesia (Coagulopathy, increased intracranial pressure, or local skin infection).
  * Patients with cardiac morbidities.
  * hypertensive disorders of pregnancy as pre-eclampsia.
  * peripartum bleeding.
  * Patients with respiratory morbidities.
  * Convulsions.
  * Bleeding diathesis.
  * Known allergy to any drugs used in this study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
frequency of Postoperative Nausea and vomiting | 24 hours
  number of patients who will have Postoperative Nausea and vomiting

SECONDARY OUTCOMES:
total amount of postoperative antiemetic consumption | 24 hours
  total amount of postoperative antiemetic consumption

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aouad MT, Yazbeck-Karam VG, Nasr VG, El-Khatib MF, Kanazi GE, Bleik JH. A single dose of propofol at the end of surgery for the prevention of emergence agitation in children undergoing strabismus surgery during sevoflurane anesthesia. Anesthesiology. 2007 Nov;107(5):733-8. doi: 10.1097/01.anes.0000287009.46896.a7. PMID 18073548
- [Background] Wang L, Huang J, Hu H, Chang X, Xia F. Commonly used antiemetics for prophylaxis of postoperative nausea and vomiting after Caesarean delivery with neuraxial morphine: a network meta-analysis. Br J Anaesth. 2024 Jun;132(6):1274-1284. doi: 10.1016/j.bja.2024.03.010. Epub 2024 Apr 15. PMID 38627136
- [Background] Yurashevich M, Habib AS. Monitoring, prevention and treatment of side effects of long-acting neuraxial opioids for post-cesarean analgesia. Int J Obstet Anesth. 2019 Aug;39:117-128. doi: 10.1016/j.ijoa.2019.03.010. Epub 2019 Apr 26. PMID 31202588
- [Background] Roofthooft E, Joshi GP, Rawal N, Van de Velde M; PROSPECT Working Group* of the European Society of Regional Anaesthesia and Pain Therapy and supported by the Obstetric Anaesthetists' Association. PROSPECT guideline for elective caesarean section: updated systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 May;76(5):665-680. doi: 10.1111/anae.15339. Epub 2020 Dec 28. PMID 33370462